CLINICAL TRIAL: NCT03905096
Title: A Study to Investigate the Effects of Donepezil on the Pharmacokinetics of BI 425809 and Vice Versa in Healthy Male and Female Subjects (Open-label, Two-treatment, Two-period, One Fixed Sequence Cross-over Design)
Brief Title: A Study in Healthy Men and Women to Test Which Effects Donepezil and BI 425809 Have on Each Other
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1346.29; 2018-004806-24 (EudraCT Number)
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: BI 425809; Drug: Donepezil
- Part 2 (Experimental)
  Interventions: Drug: BI 425809; Drug: Donepezil

INTERVENTIONS:
Drug: BI 425809 — Film coated tablet
Drug: Donepezil — Film coated tablet

SUMMARY:
The main objective of Part 1of this trial is to investigate the effect of co-administration of multiple doses of donepezil on the single-dose pharmacokinetics of BI 425809 in healthy subjects. In Part 2 the main objective is the investigation of the effect of co-administration of multiple doses of BI 425809 on the single-dose pharmacokinetics of donepezil in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12- lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria from the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception that does not contain hormones, i.e. non-hormonal intrauterine device plus condom
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open-label, two-treatment, two-period, one fixed sequence cross-over design study in order to investigate the effects of donepezil (Don) on the pharmacokinetics (PK) of BI 425809 (trial part 1) and vice versa (trial part 2) in healthy male and female subjects over a period up to 57 days in part 1 and up to 55 days in part 2.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Trial Part 1: BI 425809 / Donepezil + BI 425809: All participants were orally administered a single dose of BI 425809, 25 milligrams (mg) film-coated tablet on day 1 of visit 2 (Treatment A, Reference 1) and on day 22 of visit 3, together with multiple doses of donepezil, film-coated tablets, 5 mg once a day (qd) (1 tablet) on day 1 to 7 of visit 3 and 10 mg qd (2 tablets) on day 8 to 28 of visit 3 (Treatment B, Test 1) in the fasted state with about 240 milliliters (ml) of fluid.
- Trial Part 2: Donepezil / BI 425809 + Donepezil: All participants were orally administered a single dose of donepezil, 10 mg film-coated tablet on day 1 of visit 2 (Treatment C, Reference 2) and on day 10 of visit 3, together with multiple doses of BI 425809, film-coated tablets, 25 mg qd (1 tablet) on day 1 to 24 of visit 3 (Treatment D, Test 2) in the fasted state with about 240 milliliters (ml) of fluid.
Period: Period 1 for Trial Part 1 and 2
Arm/Group | Trial Part 1: BI 425809 / Donepezil + BI 425809 | Trial Part 2: Donepezil / BI 425809 + Donepezil
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0
Period: Period 2 for Trial Part 1 and 2
Arm/Group | Trial Part 1: BI 425809 / Donepezil + BI 425809 | Trial Part 2: Donepezil / BI 425809 + Donepezil
Started | 18 | 14
Completed | 17 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trial Part 1: BI 425809 / Donepezil + BI 425809 | Trial Part 2: Donepezil / BI 425809 + Donepezil | Total
Number analyzed (Participants) | 18 | 14 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (8.0) | 35.9 (8.6) | 37.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 21
  Male | 2 | 9 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 14 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 425809 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  For BI 425809 alone (Part 1: Treatment A, Reference 1) and BI 425809 + donepezil (Part 1: Treatment B, Test 1) plasma concentrations of BI 425809 were measured within 2 hours (h) before and at 30 minutes (min), 1 h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h, 96h, 120h, 144h, 168h after administration of BI 425809 alone or in combination with donepezil.
Time Frame: Detailed time frame is in the description section
Population: Pharmacokinetic parameter analysis set (PKS): The PKS included all subjects in the treated set (TS) who provided at least 1 pharmacokinetic (PK) endpoint that had been defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: nanomoles * hours per liter
Groups:
- BI 425809 Alone Group (Part 1: Treatment A, Reference 1): All participants were orally administered a single dose of BI 425809, 25 milligrams (mg) film-coated tablet on day 1 of visit 2 in the fasted state with about 240 milliliters (ml) of fluid (Treatment A, Reference 1).
- BI 425809 + Don Group (Part 1: Treatment B, Test 1): All participants were orally administered a single dose of BI 425809, 25 mg, film-coated tablet, on day 22 of visit 3, together with multiple doses of donepezil, film-coated tablets, 5 mg (1 tablet) once a day (qd) on day 1 to 7 and 10 mg (2 tablets) qd on day 8 to 29 of visit 3 in the fasted state with about 240 ml of fluid (Treatment B, Test 1).
Arm/Group | BI 425809 Alone Group (Part 1: Treatment A, Reference 1) | BI 425809 + Don Group (Part 1: Treatment B, Test 1)
Number analyzed (Participants) | 17 | 15
nanomoles * hours per liter | 11815.37 (1.10) | 10944.06 (1.10)
Statistical Analysis 1: Comparison: BI 425809 Alone Group (Part 1: Treatment A, Reference 1) vs BI 425809 + Don Group (Part 1: Treatment B, Test 1); Test type: Other — Relative bioavailability; ANOVA; The statistical model was analysis of variance (ANOVA) on the logarithmic scale considering the effects "subjects" as random and "treatment" as fixed; Ratio of the geometric means (T/R) % = 92.63, 90% CI 2-sided [85.34 to 100.53], Standard Deviation 12.4 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

2. Primary Outcome: Area Under the Concentration-time Curve of Donepezil in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of donepezil in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  For donepezil alone (Part 2: Treatment C, Reference 2) and donepezil + BI 425809 (Part 2: Treatment D, Test 2) concentrations of donepezil were measured within 2 hours (h) before and at 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h, 24h, 48h, 72h, 96h, 120h, 144h, 168h, 192h, 216h, 240h, 264h, 288h, 312h, 336h, after administration of donepezil alone or in combination with BI 425809.
Time Frame: Detailed time frame is in the description section
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanograms * hours per milliliter
Groups:
- Don Alone Group (Part 2: Treatment C, Reference 2): All participants were orally administered a single dose of donepezil, 10 milligrams (mg) film-coated tablet on day 1 of visit 2 in the fasted state with about 240 milliliters (ml) of fluid (Treatment C, Reference 2).
- Don + BI 425809 Group (Part 2: Treatment D, Test 2): All participants were orally administered a single dose of donepezil, 10 mg, film-coated tablet, on day 10 of visit 3, together with multiple doses of BI 425809, film-coated tablets, 25 mg qd on day 1 to 24 of visit 3 in the fasted state with about 240 ml of fluid (Treatment D, Test 2).
Arm/Group | Don Alone Group (Part 2: Treatment C, Reference 2) | Don + BI 425809 Group (Part 2: Treatment D, Test 2)
Number analyzed (Participants) | 10 | 12
nanograms * hours per milliliter | 647.16 (1.09) | 638.38 (1.09)
Statistical Analysis 1: Comparison: Don Alone Group (Part 2: Treatment C, Reference 2) vs Don + BI 425809 Group (Part 2: Treatment D, Test 2); Test type: Other — Relative bioavailability; ANOVA; The statistical model was ANOVA on the logarithmic scale considering the effect "subjects" as random and the effect "treatment" as fixed; Ratio of the geometric means (T/R) % = 98.64, 90% CI 2-sided [93.21 to 104.39], Standard Deviation 6.9 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

3. Primary Outcome: Maximum Measured Concentration of BI 425809 in Plasma (Cmax)
Description: Maximum measured concentration of BI 425809 in plasma (Cmax). For BI 425809 alone (Part 1: Treatment A, Reference 1) and BI 425809 + donepezil (Part 1: Treatment B, Test 1) concentrations of BI 425809 were measured within 2 hours (h) before and at 30 minutes (min), 1 h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h, 96h, 120h, 144h, 168h after administration of BI 425809 alone or in combination with donepezil.
Time Frame: Detailed time frame is in the description section
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomoles per liter
Groups:
- BI 425809 + Don Group (Part 1: Treatment B, Test 1): All participants were orally administered a single dose of BI 425809, 25 mg, film-coated tablet, on day 22 of visit 3, together with multiple doses of donepezil, film-coated tablets, 5 mg (1 tablet) qd on day 1 to 7 and 10 mg (2 tablets) qd on day 8 to 29 of visit 3 in the fasted state with about 240 ml of fluid (Treatment B, Test 1).
Arm/Group | BI 425809 Alone Group (Part 1: Treatment A, Reference 1) | BI 425809 + Don Group (Part 1: Treatment B, Test 1)
Number analyzed (Participants) | 17 | 15
nanomoles per liter | 293.97 (1.07) | 289.51 (1.08)
Statistical Analysis 1: Comparison: BI 425809 Alone Group (Part 1: Treatment A, Reference 1) vs BI 425809 + Don Group (Part 1: Treatment B, Test 1); Test type: Other — Relative bioavailability; ANOVA; [statistical method as in outcome 2, analysis 1]; Ratio of the geometric means (T/R) % = 98.48, 90% CI 2-sided [90.74 to 106.88], Standard Deviation 12.4 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

4. Primary Outcome: Maximum Measured Concentration of Donepezil in Plasma (Cmax)
Description: Maximum measured concentration of donepezil in plasma (Cmax). For donepezil alone (Part 2: Treatment C, Reference 2) and donepezil + BI 425809 (Part 2: Treatment D, Test 2) concentrations of donepezil were measured withing 2 hours (h) before and at 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h, 24h, 48h, 72h, 96h, 120h, 144h, 168h, 192h, 216h, 240h, 264h, 288h, 312h, 336h, after administration of donepezil alone or in combination with BI 425809.
Time Frame: Detailed time frame is in the description section
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanograms per milliliter
Arm/Group | Don Alone Group (Part 2: Treatment C, Reference 2) | Don + BI 425809 Group (Part 2: Treatment D, Test 2)
Number analyzed (Participants) | 10 | 12
nanograms per milliliter | 15.94 (1.12) | 15.96 (1.12)
Statistical Analysis 1: Comparison: Don Alone Group (Part 2: Treatment C, Reference 2) vs Don + BI 425809 Group (Part 2: Treatment D, Test 2); Test type: Other — Relative bioavailability; ANOVA; [statistical method as in outcome 2, analysis 1]; Ratio of the geometric means (T/R) % = 100.15, 90% CI 2-sided [89.01 to 112.68], Standard Deviation 14.4 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 425809 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  For BI 425809 alone (Part 1: Treatment A, Reference 1) and BI 425809 + donepezil (Part 1: Treatment B, Test 1) concentrations of BI 425809 were measured within 2 hours (h) before and at 30 minutes (min), 1 h, 2h, 3h, 3h 30min, 4h, 4h 30min, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h, 96h, 120h, 144h, 168h after administration of BI 425809 alone or in combination with donepezil.
Time Frame: Detailed time frame is in the description section
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomoles * hours per liter
Arm/Group | BI 425809 Alone Group (Part 1: Treatment A, Reference 1) | BI 425809 + Don Group (Part 1: Treatment B, Test 1)
Number analyzed (Participants) | 17 | 15
nanomoles * hours per liter | 10638.64 (1.08) | 10082.12 (1.08)
Statistical Analysis 1: Comparison: BI 425809 Alone Group (Part 1: Treatment A, Reference 1) vs BI 425809 + Don Group (Part 1: Treatment B, Test 1); Test type: Other — Relative bioavailability; ANOVA; [statistical method as in outcome 2, analysis 1]; Ratio of the geometric means (T/R) % = 94.77, 90% CI 2-sided [88.36 to 101.64], Standard Deviation 10.6 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

6. Secondary Outcome: Area Under the Concentration-time Curve of Donepezil in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of donepezil in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  For donepezil alone (Part 2: Treatment C, Reference 2) and donepezil + BI 425809 (Part 2: Treatment D, Test 2) concentrations of donepezil were measured within 2 hours (h) before and at 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h, 24h, 48h, 72h, 96h, 120h, 144h, 168h, 192h, 216h, 240h, 264h, 288h, 312h, 336h, after administration of donepezil alone or in combination with BI 425809.
Time Frame: Detailed time frame is in the description section
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanograms * hours per milliliter
Arm/Group | Don Alone Group (Part 2: Treatment C, Reference 2) | Don + BI 425809 Group (Part 2: Treatment D, Test 2)
Number analyzed (Participants) | 10 | 12
nanograms * hours per milliliter | 600.86 (1.10) | 601.20 (1.10)
Statistical Analysis 1: Comparison: Don Alone Group (Part 2: Treatment C, Reference 2) vs Don + BI 425809 Group (Part 2: Treatment D, Test 2); Test type: Other — Relative bioavailability; ANOVA; [statistical method as in outcome 2, analysis 1]; Ratio of the geometric means (T/R) % = 100.06, 90% CI 2-sided [94.56 to 105.87], Standard Deviation 6.9 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

ADVERSE EVENTS:
Time Frame: The adverse events collection time frame for BI 425809 part 1 is 8 days, for donepezil part 1 it is 28 days, and for donepezil + BI 425809 part 1 it is 14 days. The adverse events collection time frame for donepezil part 2 is 15 days, for BI 425809 part 2 it is 19 days, and for BI 425809 + donepezil part 2 it is 15 days.
Description: Treated set (TS): The TS included all subjects who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses.
Groups:
- Donepezil Group (Part 1: Treatment B, Test 1): All participants were orally administered multiple doses of donepezil, film-coated tablets, 5 mg (1 tablet) qd on day 1 to 7 and 10 mg (2 tablets) qd on day 8 to 29 of visit 3 in the fasted state with about 240 ml of fluid (Treatment B, Test 1).
- BI 425809 + Donepezil Group (Part 1: Treatment B, Test 1): All participants were orally administered a single dose of BI 425809, 25 mg, film-coated tablet, on day 22 of visit 3, together with multiple doses of donepezil, film-coated tablets, 5 mg (1 tablet) qd on day 1 to 7 and 10 mg (2 tablets) qd on day 8 to 29 of visit 3 in the fasted state with about 240 ml of fluid (Treatment B, Test 1).
- Donepezil Alone Group (Part 2: Treatment C, Reference 2): All participants were orally administered a single dose of donepezil, 10 milligrams (mg) film-coated tablet on day 1 of visit 2 in the fasted state with about 240 milliliters (ml) of fluid (Treatment C, Reference 2).
- BI 425809 Group (Part 2: Treatment D, Test 2): All participants were orally administered multiple doses of BI 425809, film-coated tablets, 25 mg qd on day 1 to 24 of visit 3 in the fasted state with about 240 ml of fluid (Treatment D, Test 2).
- Donepezil + BI 425809 Group (Part 2: Treatment D, Test 2): All participants were orally administered a single dose of donepezil, 10 mg, film-coated tablet, on day 10 of visit 3, together with multiple doses of BI 425809, film-coated tablets, 25 mg qd on day 1 to 24 of visit 3 in the fasted state with about 240 ml of fluid (Treatment D, Test 2).
Arm/Group | BI 425809 Alone Group (Part 1: Treatment A, Reference 1) | Donepezil Group (Part 1: Treatment B, Test 1) | BI 425809 + Donepezil Group (Part 1: Treatment B, Test 1) | Donepezil Alone Group (Part 2: Treatment C, Reference 2) | BI 425809 Group (Part 2: Treatment D, Test 2) | Donepezil + BI 425809 Group (Part 2: Treatment D, Test 2)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/18 | 15/18 | 13/18 | 7/14 | 4/14 | 10/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 425809 Alone Group (Part 1: Treatment A, Reference 1) (N=18) | Donepezil Group (Part 1: Treatment B, Test 1) (N=18) | BI 425809 + Donepezil Group (Part 1: Treatment B, Test 1) (N=18) | Donepezil Alone Group (Part 2: Treatment C, Reference 2) (N=14) | BI 425809 Group (Part 2: Treatment D, Test 2) (N=14) | Donepezil + BI 425809 Group (Part 2: Treatment D, Test 2) (N=14)
Dizziness (Nervous system disorders) | 2 | 6 | 5 | 2 | 1 | 6
Headache (Nervous system disorders) | 3 | 5 | 4 | 2 | 1 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 9 | 5 | 3 | 0 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 5 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 3 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 1 | 2 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03905096/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03905096/SAP_001.pdf